CLINICAL TRIAL: NCT04403542
Title: Pilot Clinical Performance of a Silicone Hydrogel Lens for Up to Six Nights of Extended Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLY935-C008
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Results first posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Refractive Errors; Myopia; Hyperopia
Keywords: Extended Wear; Contact Lens; Overnight Wear; Vision Correction; Contralateral Wear
MeSH Terms: conditions — Refractive Errors; Myopia; Hyperopia

STUDY DESIGN:
Intervention Model Description: In this contralateral study, subjects will be randomized to wear the investigational lens in 1 eye and the control lens in the other eye.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- LID018869 (OD) / Biofinity (OS) (Experimental): Lehfilcon A contact lens worn in the right eye, with comfilcon A contact lens worn in the left eye, as randomized, for approximately 1 week of continuous wear
  Interventions: Device: Lehfilcon A contact lens; Device: Comfilcon A contact lens
- Biofinity (OD) / LID018869 (OS) (Active Comparator): Comfilcon A contact lens worn in the right eye, with lehfilcon A contact lens worn in the left eye, as randomized, for approximately 1 week of continuous wear
  Interventions: Device: Lehfilcon A contact lens; Device: Comfilcon A contact lens

INTERVENTIONS:
Device: Lehfilcon A contact lens — Investigational silicone hydrogel contact lens
  Other Names: LID018869
Device: Comfilcon A contact lens — Commercially available silicone hydrogel contact lens
  Other Names: Biofinity

SUMMARY:
The purpose of this clinical study is to evaluate the on-eye performance of an investigational soft contact lens compared to a commercially available soft contact lens when worn continuously for up to 1 week.

DETAILED DESCRIPTION:
Subjects will be randomized to wear the investigational contact lens in 1 eye and the commercially available contact lens in the other eye. Subjects will be expected to attend 3 scheduled study visits: Day 1 Screening/Baseline/Dispense; Day 2 Follow-up within 4 hours of awakening (after the first night of sleeping); and Week 1 Follow-up/Exit. The expected duration of exposure to each of the study lenses for all randomized, completed subjects was approximately 7 days / 6 nights of wear.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and sign an IRB/IEC approved Informed Consent form.
* Successful wear of spherical soft contact lenses in both eyes during the past 3 months for a minimum of 5 days/week and in an extended wear modality at least 1 night/week.
* Best corrected visual acuity of 20/25 or better in each eye.
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Any condition, use of medications, or surgery that could contraindicate contact lens wear, as determined by the Investigator.
* Any habitual wear of Biofinity contact lenses.
* Pregnant or breast-feeding.
* Other protocol specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CDMA Project Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (3):
- United States (3):
  - Alcon Investigator 6402, Medina, Minnesota
  - Alcon Investigator 8046, Granville, Ohio
  - Alcon Investigator 2786, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 3 investigative sites located in the United States.
Pre-assignment Details: This reporting group includes all enrolled subjects.
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | LID018869 (OD) / Biofinity (OS) | Biofinity (OD) / LID018869 (OS)
Started | 18; 36 eyes | 18; 36 eyes
Completed | 18; 36 eyes | 18; 36 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All eyes exposed any study lens on a treatment-emergent basis
Groups:
- Total: Total of all reporting groups
Arm/Group | LID018869 (OD) / Biofinity (OS) | Biofinity (OD) / LID018869 (OS) | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (7.9) | 33.9 (10.5) | 33.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 18 | 16 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 13 | 15 | 28
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Distance Visual Acuity (VA) With Study Lenses
Description: Visual acuity (VA) was assessed for each eye individually with study lenses in place at a distance of 6 meters using a letter chart. VA was collected in Snellen and converted to logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with a lower logMAR value indicating better visual acuity. No formal hypothesis testing was planned.
Time Frame: Day 1 Dispense; Day 2 Follow-up (within 4 hours of awakening); Week 1 Follow-up/Exit
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Groups:
- LID018869: Lehfilcon A contact lens worn in the right eye or left eye, as randomized, for approximately 1 week of continuous wear
- Biofinity: Comfilcon A contact lens worn in the right eye or left eye, as randomized, for approximately 1 week of continuous wear
Arm/Group | LID018869 | Biofinity
Number analyzed (Participants) | 36 | 36
Number analyzed (eyes) | 36 | 36
logMAR
  Day 1 Dispense | -0.03 (0.05) | -0.04 (0.06)
  Day 2 Follow-up | -0.03 (0.05) | -0.03 (0.05)
  Week 1 Follow-up/Exit | -0.03 (0.05) | -0.03 (0.05)

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, approximately 7 days.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of participants. The safety analysis set includes all eyes exposed to a study lens evaluated in this study.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses
- LID018869 Ocular: Events reported in this group occurred while exposed to the lehfilcon A contact lenses
- Biofinity Ocular: Events reported in this group occurred while exposed to the comfilcon A contact lenses
- Nonocular/Systemic: Events reported in this group occurred while exposed to the study contact lenses
Arm/Group | Pretreatment | LID018869 Ocular | Biofinity Ocular | Nonocular/Systemic
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT04403542/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT04403542/SAP_001.pdf